CLINICAL TRIAL: NCT03155295
Title: Patient-specific Simulated Procedure Rehearsal for Minimally Invasive Surgery
Brief Title: Simulated Surgery Rehearsal (MIPN)
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Ahmed Ghazi, Assistant Professor, University of Rochester
Other Study IDs: 67280
Record Dates: First submitted 2017-05-10; First posted 2017-05-16 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Nephrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physical reality simulation (rehearsal): Using 3-D printing and polymer technology, the investigators will construct patient specific simulated hydrogel models designed from patients' imaging, incorporating the necessary anatomy, physiology and pathology specific to each patient. Participants with patients assigned to preoperative rehearsal will undergo pre-operative simulation only once.
  Interventions: Other: Physical reality simulation
- Virtual reality simulation: The DaVinci surgical skills simulator (DVSSS) uses a virtual reality surgical simulation platform that encompasses a variety of basic exercises specifically designed to give users the opportunity to improve their proficiency with the da Vinci surgeon console controls and basic robotic surgical skills. Participants with patients assigned to preoperative simulation will complete a refresher module on the Virtual reality simulator.
  Interventions: Other: Virtual reality simulation

INTERVENTIONS:
Other: Physical reality simulation — Using 3-D printing and polymer technology, the investigators will construct patient specific simulated hydrogel models designed from patients' imaging, incorporating the necessary anatomy, physiology and pathology specific to each patient. These models are constructed at the Laboratory for Simulation-based Translational Research at the Department of Urology. Group 1 urologists will rehearse the minimally-invasive partial nephrectomy (MIPN) surgery using these patient-specific models.
  Groups: Physical reality simulation (rehearsal)
Other: Virtual reality simulation — The DaVinci surgical skills simulator system uses a virtual reality surgical simulation platform that encompasses a variety of basic exercises specifically designed to give users the opportunity to improve their proficiency with the da Vinci surgeon console controls and basic robotic surgical skills. All urologists have already completed a basic robotic skills curriculum. Group 2 urologists will complete a refresher module on the virtual reality simulator.
  Groups: Virtual reality simulation

SUMMARY:
The purpose of the study is to evaluate patient-specific surgical simulation by permitting pre-operative rehearsals, in the form of the surgeon completing a dry run of the procedure on a model constructed from the patient's radiological studies that replicates every aspect of their organs. The investigators' aim is to evaluate the effectiveness of this form of practice in optimizing intraoperative and postoperative outcomes . The investigators hope eventually to use these rehearsals as a standard study tool for surgical training.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled to undergo MIPN surgery at the University of Rochester Medical Center
* Ability to give informed consent
* Willing to participate in the study
* Any racial or ethnic origin

Exclusion Criteria:

* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is comprised of 100 minimally invasive partial nephrectomy (MIPN) patients), 5 faculty expert urologists, and 5 trainees including four urology residents and one endourology fellow.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Warm ischemia time measured during minimal invasive partial nephrectomy surgery | At the end of each surgical procedure, approximately 24 hours after surgery
  Warm ischemia time is reported on completion of minimal invasive partial nephrectomy surgery, the metric will be measured in minutes as a continuous variable.
Estimated blood loss measured during minimal invasive partial nephrectomy surgery | At the end of each surgical procedure, approximately 24 hours after surgery
  Estimated blood loss is reported on completion of minimal invasive partial nephrectomy surgery, it is estimated by the volume of fluid in the suction irrigation at the end of surgery and measured in ml as a continuous variable.
Change in postoperative renal functions | Zero at date of randomization and serial measurements at 12 hours , 1 day and 30 days after surgery
  The difference between preoperative (within a week prior to surgery) and postoperative (12 hours , 1 day and 30 days after surgery) using estimated GFR measured through serum creatinine blood test.
Surgical complications | From date of surgery up to 30 days postoperative, every complication encountered during that time will be recorded
  Intraoperative and postoperative complications will be measured and reported using the modified Clavien-Dindo classification of surgical complications (Grade 1 to 5).
Objective evaluation of surgical performance | At the end of each surgical procedure, approximately 24 hours after surgery
  All surgical cases will be recorded and reviewed by a third party online tool that specializes in evaluation of surgical performance using the GEARS (Global Evaluative Assessment of Robotic Skills) tool
Operative time measured during minimal invasive partial nephrectomy surgery | At the end of each surgical procedure, approximately 24 hours after surgery
  Operative time is reported on completion of minimal invasive partial

SECONDARY OUTCOMES:
Positive margins of the tumor specimen | From date of randomization up to 10 days after surgery
  On pathological examination the presence or absence (+/-) and length in millimeters (mm) will be measured
Change in the volume of ratio of red blood cells to total blood volume (HCT) | Zero at date of randomization and serial measurements at 12 and 24 hours after surgery
  The difference between preoperative (within a week prior to surgery) and postoperative (12 and 24 hours after surgery) using the blood test HCT.
Hospital stay | From date of admission up to 30 days after surgery
  The length of hospital stay will be measured from time of admission to day of discharge and will be reported in days
Hospital readmission | From date of surgery up to 30 days postoperative, every hospital readmission encountered during that time will be recorded
  The readmission rates of patients enrolled in the study will be measured and reported in number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ghazi, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No